CLINICAL TRIAL: NCT06955871
Title: Clinical Investigation of Bleeding Reduction Efficacy on Toothpaste Containing 1.05% Chitosan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRO-2024-11-BLD-CHT-MS
Record Dates: First submitted 2025-04-25; First posted 2025-05-02 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Bleeding Gum; Gingivitis
MeSH Terms: conditions — Gingival Hemorrhage; Gingivitis | interventions — Chitosan; Toothpastes; Bicarbonates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test (Experimental): Toothpaste containing 1.05% Chitosan, soft-bristled toothbrush
  Interventions: Other: Toothpaste containing 1.05% Chitosan
- Positive control (Active Comparator): Toothpaste containing 67% Bicarbonate, soft-bristled toothbrush
  Interventions: Other: Toothpaste with 67% bicarbonate
- Negative control (Placebo Comparator): Silica-based NaF Toothpaste, soft-bristled toothbrush
  Interventions: Other: Silica-based NaF Toothpaste

INTERVENTIONS:
Other: Toothpaste containing 1.05% Chitosan — Toothpaste containing 1.05% Chitosan
  Arms: Test
Other: Silica-based NaF Toothpaste — Silica-based NaF Toothpaste
  Arms: Negative control
Other: Toothpaste with 67% bicarbonate — Toothpaste containing 67% Bicarbonate
  Arms: Positive control

SUMMARY:
The purpose of this study is to assess the bleeding reduction efficacy of toothpaste containing 1.05% Chitosan compared to a regular fluoride toothpaste, and compared to a toothpaste containing 67% bicarbonate.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged 18-70, inclusive.
2. Availability for the duration of the study.
3. Ability to understand and willingness to read, and sign the Informed Consent Form after the nature of the study has been fully explained to them.
4. Willingness to comply with all study procedures and clinical examination schedules.
5. Good general health (absence of any condition that, in the opinion of the study examiner, might constitute a risk to the subject while participating in the study. Examples include heart problems, valve/hip replacements etc).
6. Presence of a minimum of 20 natural teeth (excluding third molars) with facial and lingual scoreable surfaces.
7. Have a mean Modified Gingival Index (Lobene) ≥ 2.5 at screening.
8. Subjects reporting bleeding while routine toothbrushing.

Exclusion Criteria:

1. Pregnant or lactating.
2. Use of tobacco products.
3. History of alcohol or drug abuse.
4. Medical condition (especially, heart or liver problems, bleeding disorders, blood dyscrasias) or any current usage of medication that the investigator considers may compromise the subject safety, as well as, the quality of the study results.
5. Medical condition which requires pre-medication prior to dental visits/procedures.
6. History of allergy to oral hygiene products.
7. Use of anti-inflammatory, immunosuppressive, antimicrobial or anticoagulant drugs or antibiotics in the 30 days prior to the start of the study and during the course of the study.
8. Ongoing use of medications known to affect the gingival tissues (i.e. calcium channel blockers, phenytoin, cyclosporine).
9. Presence of orthodontic bands or removable partial denture(s).
10. Tumor (s) of the soft or hard tissues of the oral cavity.
11. Five or more carious lesions requiring immediate restorative treatment.
12. More than 2 periodontal pockets (>4mm deep) with bleeding on probing.
13. Any gingival condition like hyperplasia or overgrowth, that would cause difficulty in clinical assessment.
14. Participation in any other clinical study with an oral care indication or test panel within 30 days prior to the start of the study.
15. Existing medical condition which prohibits the subject from not eating or drinking for periods of up to 2 hours.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2025-04-29 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-06-04 (Actual)

PRIMARY OUTCOMES:
Gingival Bleeding | From baseline to 3 days, 7 days and 14 days after baseline.
  Gingival Bleeding Index described by Saxton and van der Ouderaa (1989).
Gingivitis | Baseline, and immediately post-brushing
  Modified Gingival Index (MGI) Lobene et al (1986)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Dental Institute of Chengdu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No